CLINICAL TRIAL: NCT04934761
Title: Study on the Effect of Capacity Shock Intervention Under Goal-directed Hemodynamic Management on P-V Loop-based Myocardial Contraction and Work
Brief Title: Study on the Effect of Capacity Shock Intervention Under Goal-directed Hemodynamic Management on P-V Loop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Red Cross Hospital (Other)
Responsible Party: Principal Investigator, Liang Bing, Deputy Director of Anesthesiology Physicians, Guangzhou Red Cross Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 202103000022
Record Dates: First submitted 2021-05-25; First posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Hemodynamics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- capacity shock (Experimental): 2ml/kg succinylateol gelatin
  Interventions: Procedure: Fluid challenge strategy
- routine management (Other): conventional strategy
  Interventions: Procedure: conventional strategy

INTERVENTIONS:
Procedure: Fluid challenge strategy — Patients received 2ml/kg of succinylateol gelatin within 10 min for fluid shock therapy after grouping, taking SVV as the management target. If SVV< 13% after shock therapy, the shock therapy was stopped and the infusion was maintained with 4ml/kg/h of crystal solution. If SVV ≥ 13% and ΔSV <10%, the individual would be excluded from the experiment. If SVV ≥ 13% but ΔSV≥10%, 2ml/kg of succinylateol gelatin was given again within 10 min for liquid shock therapy until SVV<13%, and 4ml/kg/h of crystal solution was maintained after reaching the target. If SVV≥ 13% after two shock treatments, they were excluded from the experiment. We excluded patients whose intraoperative bleeding ≥400ml and operative time ≥5 hours from the group.
  Arms: capacity shock
Procedure: conventional strategy — 4ml/kg/h of crystal solution was maintained. We excluded patients whose intraoperative bleeding ≥400ml and operative time ≥5 hours from the group.
  Arms: routine management

SUMMARY:
By observing the changes of P-V loop in capacity shock intervention Under Goal-directed Hemodynamic Management in patients undergoing total knee replacement, we investigate the effect of capacity shock on cardiac contractility and work in order to seek a more effective target plan of capacity shock for intraoperative patients.

DETAILED DESCRIPTION:
Objective:By observing the changes of P-V loop in capacity shock intervention Under Goal-directed Hemodynamic Management in patients undergoing total knee replacement, we investigate the effect of capacity shock on cardiac contractility and work in order to seek a more effective target plan of capacity shock for intraoperative patients.

Methods:20 patients with total knee replacement were enrolled in this study. Capacity shock therapy was used in Group A(n=10) and conventional strategy was used in Group B (n=10). V(t) was measured and calculated using TEE and P(t) was acquired by the analysis of patients'radial artery pressure waveform. We set five time points of parameter acquisition: after grouping (T1), the first shock completion(T2), the second shock completion (T3), 1h after shock treatment (T4), and operation completion(T5). We make up the P-V loop fitting P(t) and V(t) at each time point after the calibration of cardiac cycle.

ELIGIBILITY:
Inclusion Criteria:

ASAI-II age 40- 70 weight 48 - 72 kg.

Exclusion Criteria:

Body mass index >30 or <15 kg/m2 Valve heart disease Left ventricular ejection fraction (LVEF) is less than 50% History of lung disease Preoperative arrhythmic disorder Permanent pacemaker Need for mechanical heart Support, Severe extrinsic vascular disease Valve dysfunction OED monitoring probe insertion contraindications Patients with preoperative assessments

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Ees | Baseline，After induction
  Ees（End-systole Elasticity，mmHg/ml）
Ees | Immediately after the intervention,complete of the first round of the fluid challenge
  Ees（End-systole Elasticity，mmHg/ml）
Ees | Immediately after the intervention,complete of the second round of the fluid challenge
  Arterial elasticity is an invasively determined parameter of arterial load that is inversely related to arterial compliance
Ees | 1h after the first fluid challenge
  Ees（End-systole Elasticity，mmHg/ml）
Ees | At the end of surgery
  Ees（End-systole Elasticity，mmHg/ml）
SW | Baseline，after induction
  SW（Stroke Volume，mmHg·ml）
SW | Immediately after the intervention,complete of the first round of the fluid challenge
  SW（Stroke Volume，mmHg·ml）
SW | Immediately after the intervention,complete of the second round of the fluid challenge
  SW（Stroke Volume，mmHg·ml）
SW | 1h after the first fluid challenge
  SW（Stroke Volume，mmHg·ml）
SW | At the end of surgery
  SW（Stroke Volume，mmHg·ml）
Ea | Baseline，after induction
  Ea(Arterial elasticity, mmHg·ml)
Ea | Immediately after the intervention,complete of the first round of the fluid challenge
  Ea(Arterial elasticity, mmHg·ml)
Ea | Immediately after the intervention,complete of the second round of the fluid challenge
  Ea(Arterial elasticity, mmHg·ml)
Ea | 1h after the first fluid challenge
  Ea(Arterial elasticity, mmHg·ml)
Ea | At the end of surgery
  Ea(Arterial elasticity, mmHg·ml)

CONTACTS AND LOCATIONS:
Overall Officials: Cao Yang, Study Director — Guangzhou Red Cross Hospital
Locations (1):
- Guangzhou Red cross hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No